CLINICAL TRIAL: NCT01990638
Title: Effects of Exercise Therapy on Ventricular and Endothelial Function in Patients After Coronary Artery Bypass Surgery
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 9361701193
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: coronary artery bypass graft; Diabetes mellitus, type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fasting glucose
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DM group
  Interventions: Other: exercise capacity test
- non-DM group
  Interventions: Other: exercise capacity test

INTERVENTIONS:
Other: exercise capacity test

SUMMARY:
The purpose of this study was (1) to compare the peak exercise capacity and left ventricular diastolic function between patients with and without diabetes and (2) to investigate the interrelation among peak oxygen consumption, left ventricular diastolic function, blood sugar, and lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* well-controlled diabetes
* no history of myocardial infarction
* stable post coronary artery bypass surgery for at least 3 months

Exclusion Criteria:

* heart failure,
* valvular disease,
* abnormal kidney or liver function,
* cerebrovascular disease,
* primary pulmonary disease,
* other systemic or acute illness that may impede the testing or training

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients after coronary artery bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2004-11; Primary Completion 2005-04 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
left ventricular diastolic function | 1 week
  echocardiographic parameters

SECONDARY OUTCOMES:
flow-mediated dilation | 1 week
  flow-mediated dilation on right brachial artery
exercise capacity | 1 week
  oxygen consumption

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan